CLINICAL TRIAL: NCT03777007
Title: A Rehabilitation Tool to Determine Patient's Stay in Hospital After Joint Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derek Amanatullah (Other)
Responsible Party: Sponsor-Investigator, Derek Amanatullah, Assistant Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 48386
Record Dates: First submitted 2018-12-10; First posted 2018-12-17 (Actual); Results first posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Total Joint Replacement Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Experimental (Experimental): The application used is build upon the company's category-defining, SPARTA Platform and create a platform that streamlines the performance and management of post-acute care physical therapy. The rehab tool will provide us with functional outcome score.
  Interventions: Device: SPARTA force plate

INTERVENTIONS:
Device: SPARTA force plate — The Sparta Platform includes force plate hardware coupled with Sparta Scan software that enables quick assessment of an individual's movement and balance within minutes

SUMMARY:
SPARTA force plate is used as rehabilitation tool in this study. The device is Force Plate coupled with SPARTA scan software that enables quick assessment of individual movement and balance within minutes. The magnitude as well as efficiency of force production is analyzed to determine an patient recovery graph.

DETAILED DESCRIPTION:
The investigator hope to learn co-relation between the rehab tool and clinical findings and analyse association if any. In this study, force plate is rehab tool, which will optimize care according to the patient's specific needs and provided insights to patients length of stay in the hospital. these data driven insights will be used to observe correlation between machine and clinic data

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for Primary unilateral total joint replacement
* Patient age should be more than or equal to 18 years.
* Patient must speak English

Exclusion Criteria:

* Patients undergoing bilateral primary knee replacement surgery
* Patients undergoing revision knee replacement surgery
* No uncorrectable deformity
* No deformity greater than 15 degree
* No hip arthritis
* No wheelchair dependency

Patients not willing and capable to sign the written informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek Amanatullah, M.D. PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 55 participants signed informed consent; 40 were allocated to the study arm
Groups:
- Sparta Force Plate: The Sparta platform includes force plate hardware coupled with Sparta Scan software that enables assessment of an individual's movement and balance
Period: Overall Study
Arm/Group | Sparta Force Plate
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sparta Force Plate
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.83 (9.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 0
  Unknown or Not Reported | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Length of Stay in Hospital Through Discharge
Description: Length of stay will depend on the score generated by device.
Time Frame: Up to 8 days
Population: Participants with available data are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Sparta Force Plate
Number analyzed (Participants) | 39
days | 3 [2 to 3]

2. Secondary Outcome: Gait Aid Use
Description: The gait aide use ranges in the order of decreasing performance as Nothing > Cane/Walking Sticks > crutch > walker.
Time Frame: Preoperative and month 3 post-surgery
Population: Participants with available data at each time point are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Sparta Force Plate
Number analyzed (Participants) | 40
Participants
  Preoperative: None | 37
  Preoperative: Cane/Walking Sticks | 3
  Month 3: number analyzed (Participants) | 38
  Month 3: None | 38
  Month 3: Cane/Walking Sticks | 0

3. Secondary Outcome: Knee Society Score (KSS)
Description: To assess the effectiveness of the device by calculating Knee Society Score (KSS) at 3 months following surgery. The scale ranges from 0-100 with grading as: Score 80-100 - Excellent; Score 70-79 - Good; Score 60-69 - Fair; Score below 60 - Poor.
Time Frame: Month 3 post-surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sparta Force Plate
Number analyzed (Participants) | 40
score on a scale | 90.4 (11.39)

4. Secondary Outcome: Range of Motion
Description: To assess the effectiveness of the device by calculating range of motion (extension and flexion).
  Higher extension scores and lower flexion scores represent greater flexibility.
Time Frame: Preoperative and month 3 post-surgery
Population: Participants with available data at each time point are included in the analysis.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Sparta Force Plate
Number analyzed (Participants) | 40
degrees
  Extension - preoperative | 2.4 (3.34)
  Extension - month 3 | 0.3 (1.15)
  Flexion - preoperative: number analyzed (Participants) | 37
  Flexion - preoperative | 113.9 (11.78)
  Flexion - month 3: number analyzed (Participants) | 37
  Flexion - month 3 | 116.0 (8.54)

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Sparta Force Plate
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/07/NCT03777007/Prot_000.pdf